CLINICAL TRIAL: NCT01704027
Title: Prospective Phase II Study Evaluating the Feasibility of a Conformational Pelvic and Prostatic Radiotherapy With Simultaneous Integrated Boost Modulated-intensity Arctherapy (SIB-IMAT) in Combination With Long Term Androgen Deprivation for High Risk Localized Prostate Cancer.
Brief Title: Safety Study of Pelvic and Prostatic SIB-IMRT With Long-term Androgen Deprivation for High Risk Localized Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: termination of the trial after interim analysis. the main criterion could not be reached
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-A00694-39
Record Dates: First submitted 2012-10-02; First posted 2012-10-11 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Prostate Cancer
Keywords: Localized; High risk
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiotherapy (Experimental): Patient will receive a pelvic and prostatic simultaneous integrated boost intensity-modulated arctherapy (SIB-IMAT) in combination with three years of androgen deprivation
  Interventions: Radiation: Simultaneous integrated boost intensity-modulated arctherapy; Drug: Androgen deprivation

INTERVENTIONS:
Radiation: Simultaneous integrated boost intensity-modulated arctherapy — Three dose levels will be delivered at each fraction, 5 days a week, 30 fractions :
  * Pelvis : 55,5 Gy (1,85 Gy/fr)
  * Seminal vesicles : 66 Gy (2,2 Gy/fr)
  * Prostate : 72 Gy (2,4 Gy/fr)
Drug: Androgen deprivation — Patients will received androgen deprivation for a maximum of three years. This treatment can start six months before radiotherapy and at least the day one of radiotherapy.

SUMMARY:
The purpose of this study is to evaluate the incidence of urinary and rectal acute side effects of a pelvic and prostatic intensity-modulated arctherapy with simultaneous integrated boost (SIB-IMRT)combined with long-term androgen deprivation for patients with high risk localized prostate cancer

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the prostate
2. High risk localized adenocarcinoma defined by at least one of the following criteria:

   * Clinical stage T2c, T3 or T4
   * Gleason score ≥ 8
   * Prostate-specific antigen (PSA)≥ 20 ng/ml and ≤ 100 ng/ml
3. Patient cN0, pN0 or Nx (negative lymphadenectomy or no lymphadenectomy)
4. No pelvic adenopathy ≥ 15 mm on CT or MRI,
5. Absence of bone and/or visceral metastasis
6. Androgen deprivation beginning no later than the day of radiotherapy and up to six months before irradiation
7. Absence of prior pelvic radiotherapy,
8. Absence of surgical treatment of prostate cancer except transurethral resection performed within 4 months minimum before radiotherapy,
9. Age ≥ 18 years and ≤ 85 years
10. ECOG performance status ≤ 1,
11. Estimated life expectancy > 5 years
12. Membership of a social security system,
13. Signed informed consent.

Exclusion Criteria:

1. Prostate cancer histology other than adenocarcinoma,
2. pN1 patients (lymph node dissection after histologically proven)
3. PSA > 100 ng/ml
4. History of cancer within 5 years prior to trial entry (with the exception of basal cell carcinoma skin)
5. Patient with severe hypertension uncontrolled by appropriate treatment (≥ 160 mm Hg systolic and / or ≥ 90 mm Hg diastolic)
6. Contra-indication for pelvic irradiation (eg scleroderma, chronic inflammatory disease of the digestive tract, etc ...)
7. Contra-indication to agonists or antagonists of LH-RH
8. Bilateral hip prosthesis,
9. Patients already included in another clinical trial with an experimental molecule,
10. Persons deprived of liberty or under guardianship
11. Unable to undergo medical test for geographical, social or psychological.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-10; Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Acute urinary and rectal toxicities as a Measure of treatment specific Safety and Tolerability | From start of radiotherapy to six months after the end of radiotherapy
  Acute urinary and rectal toxicities will be assessed according to the NCI CTCAE v4.0 quotation each week during radiotherapy treatment period up to six months after the end of the radiotherapy treatment period.

SECONDARY OUTCOMES:
To evaluate the late urinary and rectal toxicities | for each patient every 6 months after the end of radiotherapy up to 5 years.
Evaluate the 5-year biochemical-free survival | for each patient from zero day up to 7 day after the end of radiotherapy, 6 weeks, 3 months, and every 6 months after the end of radiotherapy up to 5 years.
Evaluate the metastase-free survival | for each patient from zero day up to 7 day after the end of radiotherapy, 6 weeks, 3 months, and every 6 months after the end of radiotherapy up to 5 years.
To evaluate the specific survival | for each patient from inclusion up to 5 years after the end of radiotherapy.
To evaluate the overall survival | for each patient from inclusion up to 5 years after the end of radiotherapy.
To evaluate the quality of life | inclusion day, from zero day up to 7 day after the end of radiotherapy, 6 weeks after the end of the radiotherapy, 3 months after the end of the radiotherapy, every 6 months after the end of radiotherapy up to 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Etienne MARTIN, MD, Principal Investigator — Centre Georges François Leclerc
Locations (1):
- Centre Georges-François Leclerc, Dijon, Burgundy, France